CLINICAL TRIAL: NCT05076123
Title: Efficacy of Modified Constraint Induced Movement Therapy Combined With Threshold Electrical Stimulation in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, research assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: doctoral thesis
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2021-09

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; Electrical stimulation; Upper extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group-1 (M-CIMT group) (Experimental): participants in this group will be trained with Modified Constraint Induced Therapy (M-CIMT) in addition to conventional therapy. M-CIMT is shorter versions of CIMT. The original CIMT devotes six or more hours for therapy and constraining of the intact arm for 90% of waking hours per day and over a period of two weeks. Researchers have observed that such a schedule of CIMT is exhaustive and possibly resulting in non-compliance. Because of this reason,s Modified shorter versions of CIMT (mCIMT) have been designed by researchers. Duration of M-CIMT interventions varies from 2 to 10 weeks and the treatment time also varies from as short as 30 minutes to three hours per day in various studies. Nevertheless both CIMT and mCIMT have shown promising success. M-CIMT emphasizes massed practice with the affected upper limb.
  Interventions: Other: Modified Constraint Induced Therapy and Threshold Electrical Stimulation
- Experimental group-2 (M-CIMT+TES group) (Experimental): participants in this group will be trained with Modified Constraint Induced Therapy (M-CIMT) and threshold electrical stimulation (TES) in addition to conventional therapy. TES is based on low-intensity (<100 Hz) and long-duration current and is applied with superficial electrodes. TES provides a natural proprioception by depolarizing the sensory and motor nerves without causing any muscle contraction. TES can improve motor learning and motor performance by improving connections between sensory-motor cortical association regions in the brain.
  Interventions: Other: Modified Constraint Induced Therapy and Threshold Electrical Stimulation
- Control group (No Intervention): participants in this group will be trained with conventional therapy. Conventional therapy consists of strength training, stretching exercises and functional activity training.

INTERVENTIONS:
Other: Modified Constraint Induced Therapy and Threshold Electrical Stimulation — M-CIMT emphasizes massed practice with the affected upper limb with restraining unaffected limb by a mitt. Threshold electrical stimulation is based on low-intensity (<100 Hz) and long-duration current and is applied with superficial electrodes.
  Arms: Experimental group-1 (M-CIMT group); Experimental group-2 (M-CIMT+TES group)

SUMMARY:
This study, it is aimed to investigate the effectiveness of applied modified constraint-induced movement therapy (MCIMT) with threshold electrical stimulation (TES) in addition to conventional therapy (therapeutic exercise program) in patients with stroke. Before and after the treatment program we will evaluate, the pain level of the participants measured with a visual pain scale; sensory functions with Semmes Weinstein monofilament test battery; muscle tone, and spasticity with the modified Tardieu scale and Digital Palpation Device, which has a very high proof value; functional status with Wolf motor function test and Motor Activity Log; quality of life will be assessed by Stroke Specific Quality of Life Scale. Participants will be included in the study according to the inclusion criteria, the first evaluation of the participants will be made according to the evaluation parameters, and the participants will be randomly distributed into three groups. The first group will be treated with M-CIMT, the second group will be treated with MCIMT with TES for 4 weeks, and the third group will be the control group. A total of 45 participants will be included in the study.

DETAILED DESCRIPTION:
This study, it is aimed to investigate the effectiveness of applied modified constraint-induced movement therapy (MCIMT) with threshold electrical stimulation (TES) in addition to conventional therapy (therapeutic exercise program) in patients with stroke. MCIMT treatment applied together with TES will be performed with electric stimulation without causing discomfort in patients with stroke and at the same time, the duration of use of the affected extremity can be extended with task-oriented exercises with MCIMT treatment. In this way, the efficiency of the applied treatment program will be evaluated, and the gains obtained will be investigated and presented as a suggestion to physiotherapists working with stroke patients. Before and after the treatment program we will evaluate, the pain level of the participants measured with a visual pain scale; sensory functions with Semmes Weinstein monofilament test battery; muscle tone, and spasticity with the modified Tardieu scale and Digital Palpation Device, which has a very high proof value; functional status with Wolf motor function test and Motor Activity Log; quality of life will be assessed by Stroke Specific Quality of Life Scale. Participants will be included in the study according to the inclusion criteria, the first evaluation of the participants will be made according to the evaluation parameters, and the participants will be randomly distributed into three groups. The first group will be treated with M-CIMT, the second group will be treated with MCIMT with TES for 4 weeks, and the third group will be the control group. A total of 45 participants will be included in the study. Participants in all three groups will be included in the routine conventional physiotherapy program. MCIMT and TES treatment will be applied three days a week for a total of four weeks. Each treatment session will continue for one and a half hours. A total of two evaluations will be applied before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients aged between 18-80 years
* Having had a stroke at least 3 months and at most 24 months ago
* Having an active range of motion of the upper extremity which is stated below:

Shoulder flexion and abduction of at least 45 degrees Starting from a 90° flexion position, at least 20° elbow extension Starting from full of wrist flexion position at least 20° wrist extension At least 10° of extension at the metacarpophalangeal and interphalangeal joints of all fingers

- Absence of severe spasticity to affect the treatment (spasticity in any joint of the upper extremity ≤2 according to the Modified Ashworth Scale)

Exclusion Criteria:

* Uncontrollable arrhythmia and/or hypertension
* Presence of advanced sensory deficit
* Visual and hearing problems
* Presence of severe spasticity to affect the treatment (spasticity in any joint of the upper extremity >2 according to the Modified Ashworth Scale)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Range of motion (ROM) of upper extremity | Change from baseline Range of Motion (ROM) at week 4.
  A universal goniometer will be used to evaluate ROM (shoulder flexion and abduction, elbow flexion and extension, wrist flexion and extension and extension of fingers). Kendall-McCreary criteria will be considered in the assessments. Measurements will be repeated three times and the average value will be used in the statistical analysis.
Pain of upper extremity | Change from baseline pain at week 4.
  Pain (pain of shoulder, elbow, wrist and fingers) will be evaulated with VAS (Visual Analog Scale). The VAS consists of a 10 cm straight line which presents a continuum of intensity and has verbal anchors at opposite ends representing 'no pain' at the bottom and 'pain as bad as it can be' at the top. The participants will be asked to mark the representing point of their pain levels. The values will be recorded in centimeters.
Muscle tone and viscoelastic properties of muscle: | Change from baseline muscle tone at week 4.
  Muscle tone will be evaluated with the Myoton®PRO Digital Palpation Device. It is an evidence-based Class 1 device that evaluates the bio-mechanical properties of soft biological tissues in a non-invasive, objective, reliable, inexpensive, quick and easy way. Myoton® PRO is used in research to evaluate superficial skeletal muscles, connective tissues such as tendons and ligaments, and other soft tissues
Severity of spasticity | Change from baseline severity of spasticity at week 4.
  The Modified Tardieu scale will be used to assess the severity of spasticity. In this method, the severity of spasticity is evaluated at different rates determined. At the joint, the first angle at which the increase in resistance is detected is recorded. The range of motion is compared to the angle at completion. The Stretching Velocities are as follows: V1: As slow as possible (slower than the gravity fall speed of the limb segment) V2: At the rate of gravity fall of the limb V3: As fast as possible (faster than the normal gravity fall speed of the limb).
Superficial sensory function | Change from baseline superficial sense of upper extremity at week 4.
  The Semmes Weinstein monofilament test battery will be used to evaluate the superficial sense of upper extremity. Monofilaments of varying thickness between 1.65 and 6.65 are used in this test battery. The evaluator applies in order from the smallest filament to the largest filament, the test is stopped when the monofilament is detected by the evaluator. It is a reliable method used in the superficial sensory evaluation of stroke patients.
Health-Related Quality Of Life | Change from baseline quality of life at week 4.
  "Stroke-specific quality of life scale (SSQOL)" will be used to evaluate quality of life. SSQOL; It is a valid and reliable scale consisting of 12 subsections, including energy, family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper extremity function, vision and productivity, and a total of 49 questions. It is graded with Likert-type scoring ranging from 1 to 5.
Functional Status | Change from baseline functional status at week 4.
  Wolf Motor Function test is used to evaluate upper extremity motor functions. For 15 activities, data is collected in 2 areas, "Functional Skill" and "Performance Time". Using the "Functional Skills Scale", each activity is evaluated between 0-5 points (0= Never used the affected hand during the activity, 5= Normal movement). The average score is calculated for the Functional Skill Scale. Performance Time" is recorded in seconds (sec).
Motor activity | change from baseline motor actvity at week 4.
  Motor activity diary-28 (MAG-28) will be used to evaluate motor activity. The MAG-28 is a valid and reliable scale designed to examine how often and how well a person uses their affected arm outside of the treatment session. It consists of two scales that question how often the patient uses the affected side upper extremity for each activity during daily activities (turning the light switch, opening the door, etc.) (Use Frequency Scale), and if so, how well he or she can perform the activity (Movement Quality Scale). The patient scores himself between 0 and 5 (0 = I do not use my affected arm at all, 5 = I use my affected arm with the same frequency/quality as before the stroke). For the average score, the total scores of both scales are calculated separately and divided by the number of questions

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Mete, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No